CLINICAL TRIAL: NCT03305302
Title: Isolation and Establishment of Gustatory Cell Lines in Patients Operated on for Cancer of the Mobile Tongue - ImmortTasteCELL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ZWETYENGA 2017
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cancer of the Tongue
MeSH Terms: conditions — Tongue Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sample of cancerous epithelium from the tongue — Harvesting and culture of cancerous epithelium from the surgical piece

SUMMARY:
In terms of incidence, cancer of the tongue is one of the leading cancers in France. Moreover, this cancer is associated with physiological complications ranging from swallowing disorders to loss of taste. Following surgery, impaired perception of food taste may lead to cachexia. It is therefore necessary to carry out research in the field of impaired taste, notably with regard to the regeneration of taste buds. However, there is currently no available functional model of taste bud cells.

It is therefore necessary to obtain a cell line of human taste cells. These immortalised human cells will allow us to better orient our investigations for applications in humans: search for and characterisation of "taste modifiers" synthesised using organic chemistry, able to trigger the perception of food in cases of taste loss or taste impairment.

Moreover, given recent studies conducted by the investigating team proposing the existence of a fatty taste and its implication in obesity, the work of the team could be oriented towards the synthesis of lipid-receptor agonists, by analogy with artificial sweeteners instead of sugar. The availability of these chemical molecules would lead to a reduction in lipid intake as these agents contain no (or very few) calories. They will act as an organoleptic decoy.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 70 years old,
* with cancer of the mobile tongue
* requiring surgery

Exclusion Criteria:

- chronic smokers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Immortalised human taste bud cells, isolated from the fungiform tastebuds of patients with cancer of the mobile tongue. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France